CLINICAL TRIAL: NCT03709641
Title: A Single-Arm, Single-Center, Randomized, Single-Masked Study to Evaluate Restylane Defyne for Canalicular Occlusion in Participants With Mild to Moderate Dry Eye Disease
Brief Title: A Study to Evaluate the Safety and Effectiveness of Restylane-Defyne for Punctual Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John C Meyer, MD (Other)
Responsible Party: Sponsor-Investigator, John C Meyer, MD, Ophthalmologist, The Eye Care Institute
Organization: The Eye Care Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0918
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Mild to Moderate Dry Eye Disease
Keywords: Dry Eye Disease; Restyalne Defyne
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Study is set as a single-arm, randomized, single-masked to evaluate Restylane Defyne for canalicular occlusion in participants with mild to moderate dry eye disease. Each participant will have a screening visit, it is then participants will be provided with informed consent form to review and ask questions before written informed consent is obtained. Screening visit occurs 30 days prior to 42 days and will be seen for follow-up exams at 3 , 14 and 42 days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Restylane Defyne receiver (Experimental): Participants will receive Restyane Defyne injected into punctum of one eye.
  Interventions: Device: Restylane Defyne

INTERVENTIONS:
Device: Restylane Defyne — Restylane is a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL

SUMMARY:
A study which participants with mild to moderate dry eye disease will have a punctum of one eye injected with Restyalne Defyne and the other eye injected with saline solution. Participants will be evaluated over four visits.

ELIGIBILITY:
Inclusion Criteria:

* Twenty-one (21) to 80 years of age
* Baseline Ocular Surface Disease Index score of at least 13 with no more than 3 responses of "not applicable" for each eye individually
* In the study eye, a baseline Schirmer test with anesthetic of ≤ 10 mm/5 minute
* Literate, able to speak English and able to complete the questionnaire independently
* Willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol.

Exclusion Criteria:

* Use of ophthalmic cyclosporine or lifitegrast within 30 days prior to Day 0.
* History of surgical punctal occlusion (e.g., cautery), canalicular infection or canalicular surgery.
* Corneal transplant in either eye
* Ocular surgery (such as cataract surgery or LASIK) in either eye within six months of the Baseline Visit.
* A systemic condition or disease not stabilized or judged by the investigator to be incompatible with participation in the study (e.g. current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease).
* The history or presence of any ocular disorder or condition in either eye that, in the opinion of the investigator, would interfere with the interpretation of the study results (e.g., significant corneal or conjunctival scarring, pterygium or nodular pinguecula; current ocular infection (except mild blepharitis), conjunctivitis or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; history of ocular herpetic infection; evidence of keratoconus; lid or lacrimal cancer.
* Active severe systemic allergy, seasonal allergies, rhinitis or sinusitis requiring treatment (i.e. antihistamines, decongestants, oral or aerosol steroids).
* Use of steroids, including administration by systemic, inhaled or topical ocular routes (dermatologic steroids not applied to the eyelids are allowed).
* Participation in a clinical trial during the past 30 days
* Women who are pregnant, planning a pregnancy, or nursing at study entry

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Evaluating change in Schirmer score from baseline | 42 days after screening visit
  Maximum length of tears absorbed on test strips recorded.

SECONDARY OUTCOMES:
Evaluating change in Ocular Surface Disease index (OSDI) score from baseline | 42 days after screening visit
  Participants answer 12 question questionnaire. Scores from section I,II, and III
Evaluating change in corneal staining score from baseline. | 42 days after screening visit
  1.0mg sodium fluorescein strips on lower eye lids for one minute. 5 corneal regions graded using cobalt filter to maximized view of fluorescence.
Evaluating Tear break-up time (TBUT) from baseline. | 42 days after screening visit
  Performed by Keratograph 5M per manufacturer's directions.
Evaluating tear meniscus height from baseline. | 42 days after screening visit.
  Performed by Keratograph 5M per manufacturer's directions.

CONTACTS AND LOCATIONS:
Overall Officials: John C Meyer, MD, Principal Investigator — The Eye Care Institute
Locations (1):
- The Eye Care Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03709641/Prot_000.pdf